CLINICAL TRIAL: NCT04592055
Title: The Effect of COVID-19 on the Glycemic Control in Patients With Diabetes Mellitus
Brief Title: The Effect of COVID-19 on Diabetes Mellitus
Acronym: COVID-19-DM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uşak University (Other)
Responsible Party: Sponsor
Other Study IDs: UU-DM002
Record Dates: First submitted 2020-10-16; First posted 2020-10-19 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Diabetes Mellitus; Covid19
MeSH Terms: conditions — Diabetes Mellitus; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aimed to evaluate the effect of SARS-COV-2 infection on metabolic status in patients with diabetes mellitus. Patients' HbA1c levels before and after SARS-COV-2 infection will be evaluated.

DETAILED DESCRIPTION:
In this time pediods, all patients with RT-PCR positive for SARS-COV-2 will be analysed for the presence of diabetes mellitus. Previous HbA1c levels will be obtained from hospital records. In these patients, previous A1c levels and A1c levels 3 months after the SARS-COV-2 infection will be compared.

ELIGIBILITY:
Inclusion Criteria:

- All hospitalised diabetic patients with RT-PCR- positive for SARS-COV-2 will be enrolled.

Exclusion Criteria:

- The absence of diabetes mellitus RT-PCR- negative for SARS-COV-2 Non-hospitalised patients

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All hospitalised diabetic patients with RT-PCR- positive for SARS-COV-2 will be enrolled and evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
A1c | 6 months (3 months before and after COVID-19
  the change in A1c levels

CONTACTS AND LOCATIONS:
Overall Officials: Cevdet Duran, Prof, Principal Investigator — Uşak University
Locations (1):
- Usak University Training and Research Hospital, Uşak, Turkey (Türkiye)